CLINICAL TRIAL: NCT05834686
Title: An Exploratory Clinical Study of HER2 Expression of Circulating Tumor Cells : Predictive and Prognostic Value in HER2-positive Advanced Breast Cancer Patients Treated With ADC
Brief Title: HER2 Expression of CTC to Predict Response in HER2-positive Advanced Breast Cancer Patients Treated With ADC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Breast-CTC-HER2
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: HER2 expression of circulating tumor cells — Detect HER2 expression of circulating tumor cells dynamically during ADC-based treatment in HER2-positive ABC

SUMMARY:
To evaluate the predictive and prognostic value of HER2 expression of circulating tumor cells in HER2-positive advanced breast cancer patients treated with ADC

ELIGIBILITY:
Inclusion Criteria:

* Has pathologically documented breast cancer that:

  1. Is unresectable or metastatic
  2. has confirmed HER2-positive expression defined as IHC 2+/ISH+ or IHC 3+
  3. was previously treated with trastuzumab and taxane in the advanced setting or progressed within 6 months after neoadjuvant or adjuvant treatment involving a regimen including trastuzumab and taxane
* Has adequate cardiac, bone marrow, renal, hepatic and blood clotting functions
* Receives anti-HER2 ADC treatment
* Life expectancy > 3 months
* Evidence of measurable or evaluable disease (RECIST 1.1 criteria)in the 28 days before selection
* ECOG ≤2

Exclusion Criteria:

* Has uncontrolled or significant cardiovascular disease
* Has history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
* Has any medical history or condition that per protocol or in the opinion of the investigator is inappropriate for the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with HER2-positive breast cancer (according to International Classification of Diseases-10, ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | 3 years
  PFS was defined as the time from the start of treatment to either the first documented disease progression or death from any cause

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2years
  ORR was defined as the proportion of patients with a complete response or a partial response
Overall survival(OS) | 5 years
  OS was defined as the time from the start of treatment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, Study Director — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China